CLINICAL TRIAL: NCT01043653
Title: Assessing Recovery in Veterans With Serious Mental Illness
Brief Title: Assessing Mental Illness Recovery
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D7156-R
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Serious Mental Illness
Keywords: recovery; serious mental illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no specimens collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Maryland Assessment of Recovery in Serious Mental Illness: Individuals with serious mental illness treated in mental health outpatient programs

SUMMARY:
In 2003 the VA Undersecretary's Action Agenda mandated that mental health services throughout the system be transformed to a recovery model. That mandate and many of the Workgroup recommendations have since been formalized in the Uniform Mental Health Services Package, which specifies a range of recovery-oriented services that must be available to veterans. A key aspect of these policy mandates is the need to assess recovery status of veterans and to monitor their progress over time as a way to evaluate the effectiveness of recovery services. However, there is no established instrument that is suitable for system-wide application. The purpose of this project is to develop a reliable, valid and practical measure of recovery, and use the measure in a study to better understand recovery in individuals with serious mental illness.

DETAILED DESCRIPTION:
Mental health care in the United States and Western Europe is undergoing a seismic shift in values. The paternalistic, medical model of care that has dominated practice for more than 75-years is being challenged by an activist group of consumer-survivors, with the support of public officials and an increasing number of professionals. The centerpiece of this shift is the recovery model, which assumes that all consumers have the capacity to improve and develop a life distinct from their illness. The consumer model of recovery involves a non-linear process in which the consumer gradually adapts to, and moves beyond the illness. It emphasizes hope, empowerment, and control of one's life. This model stands in contrast to scientific and clinical models, which view recovery as an outcome, primarily involving reduced symptoms and improved functional capacity.

The public health significance of the consumer perspective is underscored by the President's New Freedom Commission on Mental Health (2003), which enunciated two guiding principles for mental health services in the US: First, services and treatments must be consumer and family centered, geared to give consumers real and meaningful choices about treatment options and providers. Second, care must focus on increasing consumers' ability to successfully cope with life's challenges, on facilitating recovery, and on building resilience, not just managing symptoms. In response to the Commission report the VA has mandated a shift to a recovery model and committed a large amount of resources to implementing it throughout the system.

Despite this political and programmatic change, there is little scientific literature on the nature of recovery or the factors that contribute to it. Systems change is being driven by social mandate and consensual agreement rather than empirical support. It is essential that the consumer model of recovery be subjected to empirical study if it is to have a meaningful and lasting impact on systems and patterns of care. It is also critical to evaluate the recovery-oriented systems of care that have been developed. Two factors that have limited empirical study of the construct and treatment programs are: a) the absence of a scientifically grounded conceptual model of recovery, and b) the lack of a reliable and valid assessment instrument to measure recovery status. The purpose of this project is to develop and evaluate a psychometrically sound assessment scale using Bandura's social cognitive theory as a conceptual model for the recovery construct.

The Specific Aims are: 1) to evaluate and refine the draft version of the Maryland Assessment of Recovery in Serious Mental Illness (MARS), 2) evaluate its test-retest reliability and validity, and 3) to examine recovery status and the relationship of recovery to hypothesized mediators and moderators over a 1-year retest interval.

ELIGIBILITY:
Inclusion Criteria:

* chart diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder I (with mania), or major depression with psychotic features, with a history of a minimum of 2 psychotic exacerbations, or Psychosis NOS
* A minimum of 2 psychotic exacerbations(confirmed by medical record, provider report, or patient self-report);
* Are receiving services from participating study sites and have had a minimum of two service visits within the last 6 months;
* Have received mental health services for a minimum of 3-years;
* Age between 25 and 65;
* Able to provide informed consent; and
* Able to complete protocol assessments (estimation from medical record and/or mental health provider that person can read at 5th grade level and sustain attention to study tasks for required period of time).

Exclusion Criteria:

* Severe or profound mental retardation as indicated by chart review

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We have elected to focus on individuals meeting accepted criteria for serious mental illness, including a diagnosis of schizophrenia or schizoaffective disorder, bipolar I disorder (with mania), and major depression with psychosis. Individuals meeting these criteria represent a large population with significant costs and health concerns for VA. Further, they are the primary target of efforts to transform mental health care in VA to a recovery model, making this an arena in particular need of a sound recovery instrument.
  We have elected to limit our sample to people in treatment for several reasons. One can surmise that most people not in treatment are new cases, very ill (e.g., homeless), or doing very well.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Bellack, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (3):
- United States (3):
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - University of Maryland, Division of Psychiatry, Baltimore, Maryland
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maryland Assessment of Recovery in Serious Mental Illness
Started | 250
Completed | 186
Not Completed | 64

BASELINE CHARACTERISTICS:
Groups:
- Maryland Assessment of Recovery in Serious Mental Illness: Individuals with serious mental illness treated in VA mental health outpatient programs
Arm/Group | Maryland Assessment of Recovery in Serious Mental Illness
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 206

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Scale (PANSS)
Description: The PANSS is a clinician-rated measure of the presence and severity of symptoms of psychosis. A total score was calculated by averaging the responses on the items (range=1 to 7) scores, with higher scores indicating greater severity of psychiatric symptoms.
Time Frame: ~1-year
Population: The PANSS had additional missing data from 3 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maryland Assessment of Recovery in Serious Mental Illness
Number analyzed (Participants) | 183
units on a scale
  Baseline | 1.9 (0.4)
  Follow-up | 1.8 (0.4)

2. Secondary Outcome: Maryland Assessment of Recovery in Serious Mental Illness
Description: The Maryland Assessment of Recovery in Serious Mental Illness is a self-report measure of recovery in people with serious mental illness. A total score was calculated by summing item responses (range=25 to 125), with higher total scores indicating greater self-reported recovery.
Time Frame: ~ 1-year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maryland Assessment of Recovery in Serious Mental Illness
Number analyzed (Participants) | 186
units on a scale
  Baseline | 95.9 (19.5)
  Follow-up | 95.7 (19.2)

ADVERSE EVENTS:
Time Frame: ~ 1 year
Arm/Group | Maryland Assessment of Recovery in Serious Mental Illness
Serious Adverse Events (participants affected / at risk) | 9/250
Other Adverse Events (participants affected / at risk) | 0/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maryland Assessment of Recovery in Serious Mental Illness (N=250)
Psychiatric Hospitalization (Psychiatric disorders) | 6 (6) — All psychiatric hospitalizations that occurred during the study were reported to the local IRB and unrelated to study participation
Medical Hospitalization (General disorders) | 3 (3) — All medical hospitalizations that occurred during the study were reported to the local IRB and unrelated to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes